CLINICAL TRIAL: NCT04373174
Title: The Effect of Regional Anesthesia Techniques on Brain Tissue Oxygenation in Thoracic Surgery Operations Where Single Lung Ventilation is Applied
Brief Title: The Effect of Regional Anesthesia Techniques on Brain Tissue Oxygenation in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BYIERH
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Thoracic Surgery; Epidural Anesthesia; Cerebral Oxygen Saturation

STUDY DESIGN:
Intervention Model Description: prospective,randomized
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): Thoracic Epidural block + Regional oximetry probe will be placed in the frontal area of the head
  Interventions: Device: Regional oximetry probe; Procedure: Thoracic Epidural block
- Group P (Sham Comparator): Regional oximetry probe will be placed in the frontal area of the head
  Interventions: Device: Regional oximetry probe

INTERVENTIONS:
Device: Regional oximetry probe — Regional oximetry probe will be placed in the frontal area of the head
Procedure: Thoracic Epidural block — Thoracic epidural block will be applied to the patients before the operation begins
  Arms: Group E

SUMMARY:
Today, it is preferred that the lung with pathology for thorax surgery is not under ventilation during operation in terms of reliability and ease of operation.

For this reason, the anesthesia approach is characteristic and it is ensured that the single lung is not ventilated during the operation by means of specially manufactured intubation tubes. This application can disrupt tissue oxygenation due to both Operation position and single lung ventilation.

Thoracic epidural analgesia, which is applied as the gold standard of Thoracic Surgery, is applied prior to the operation and is provided to assist in postoperative analgesia.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of thoracic epidural analgesia method on brain tissue oxygenation in patients with single lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* Underwent Thoracic Surgery

Exclusion Criteria:

* Local anesthetic allergy,
* Bleeding is a diathesis disorder
* Allergic to the drugs used,
* Patients who are not reluctant to participate in the study,
* Presence of infection in the block area,
* Patients whose body mass index is over 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
rso2 | peroperative 2 hours
  Regional oximetry probe will be placed in the frontal area of the head

SECONDARY OUTCOMES:
po2 | peroperative 2 hours
  Arterial blood gas oxygen pressure
ETCO2 | peroperative 2 hours
  End-tidal carbon dioxide (ETCO2) level

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Study Director — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No